CLINICAL TRIAL: NCT04450693
Title: A Multicenter Phase 3 Confirmatory Trial of Biotherapy Using Cryopreserved Human Umbilical Cord (TTAX01) for Late Stage, Complex Non-healing Diabetic Foot Ulcers (AMBULATE DFU II)
Brief Title: Cryopreserved Human Umbilical Cord (TTAX01) for Late Stage, Complex Non-healing Diabetic Foot Ulcers (AMBULATE DFU II)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioTissue Holdings, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TTAX01-CR005
Record Dates: First submitted 2020-06-25; First posted 2020-06-29 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Foot Infection; Non-healing Wound; Non-healing Diabetic Foot Ulcer
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the test article, the trial is open label, with no blinding of the site staff. The determination of wound closure will be made by the Investigator based on visual and tactile assessment of the wound. To reduce bias in the ascertainment of closure, one independent blinded reviewer will review the image obtained from a wound measurement device in each case where the Investigator makes a determination of closure. Discordant opinions will be adjudicated by a second independent blinded reviewer who will examine multiple additional images taken at various angles to the wound surface.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TTAX01 (Experimental): TTAX01 plus standard of care
  Interventions: Biological: TTAX01; Other: Standard care
- Control (Other): Standard care alone
  Interventions: Other: Standard care

INTERVENTIONS:
Biological: TTAX01 — TTAX01 is a cryopreserved human umbilical cord product derived from donated human placental tissue following healthy, live, caesarian section, full-term births after determination of donor eligibility and placenta suitability. TTAX01 is manufactured by TissueTech Inc. utilizing a proprietary CRYOTEK® process, which devitalizes the living cells but retains the natural structural and biological characteristics relevant to this tissue. TTAX01 is aseptically processed in compliance with current Good Tissue Practices (cGTP). TTAX01 will be manufactured in various sizes, stored in a medium of lactated Ringer's/glycerol (1:1).
  Arms: TTAX01
Other: Standard care — Standard care is defined in this protocol to consist of the following:
  * Debridement;
  * Wound cleansing, using sterile saline, a non-ionic cleanser or a hypochlorous solution. Antiseptic agents including hydrogen peroxide, acetic acid, chlorhexidine, povidone/iodine, and cetrimide should not be used. Topical antimicrobials and silver dressings are also prohibited;
  * Primary wound dressings including a non-adherent, standard foam pad with or without a hydrogel beneath the dressing, or and alginate dressing, as is appropriate to maintain a moist wound environment while managing exudate;
  * A secondary retention bandage appropriate to the amount of wound exudate, so as to avoid maceration of the peri-wound skin;
  * Off-loading device appropriate to the location of wound with full length boot or total contact cast (unless not appropriate where a substitute off-loading device can be made with sponsor approval); and,
  * Appropriate use of systemic antibiotics.

SUMMARY:
It is hypothesized that application at 4-week or greater intervals of the human placental umbilical cord tissue TTAX01 to the surface of a well debrided, complex diabetic foot ulcer (DFU) will, with concomitant management of infection, result in a higher rate of wounds showing complete healing within 25 weeks of initiating therapy, compared with standard care alone. This second confirmatory Phase 3 study examines a population of diabetic foot ulcer patients having adequate perfusion, with or without neuropathy, and a high suspicion of associated osteomyelitis in a complex, high grade wound.

DETAILED DESCRIPTION:
This trial is designed as a confirmatory study of the benefits and risks of TTAX01 when used in the treatment of Wagner Grades 3 and 4 DFU. Experience with the use of a cryopreserved umbilical cord (UC) product in treating such wounds, both prior to this IND and under this IND, has indicated that a frequency of application of no shorter than every 4 weeks is associated with better than expected outcomes. Although treatment cannot be blinded, a "standard care only" arm is included to control for the benefits of aggressive baseline debridement combined with aggressive (6 weeks systemic) antibiotics. Current treatment guidelines indicate that aggressive debridement plus 1-2 weeks of antibiotics, or, minor debridement plus 6 weeks of antibiotics, would produce equivalent outcomes, although the evidence is not strong. By utilizing both maximum debridement and maximum antimicrobial therapy, the standard care described in this protocol may result in healing rates somewhat superior to current standard practice.

The design of this second confirmatory study is matched to the design of the Phase 2 efficacy study TTCRNE-1501, with the exception of extending the primary endpoint from a landmark analysis at 16 to a "wound survival" analysis through 26 weeks, utilizing a proportional risk analysis rather than a simple test of proportions. This design consideration is based on analysis of previous studies (see Background section), and a desire to fold data from every visit into the primary analysis, rather than generating an excessive number of secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* The subject has signed the informed consent form
* The subject is male or female, at least 18 years of age inclusive at the date of Screening
* The subject has confirmed diagnosis of Type I or Type II diabetes
* The subject's index ulcer is located on the plantar surface, inter digital, heel, lateral or medial surface of the foot
* The subject has an index ulcer with visible margins having an area ≤ 12.0 cm2 when measured by the electronic measuring device at Screening
* The subject's index ulcer extends beyond the dermis, into subcutaneous tissue with evidence of exposed bone, tendon, muscle and/or joint capsule
* The subject presents with history, signs or symptoms leading to a clinical suspicion of osteomyelitis in the opinion of the Investigator supported by positive Probe to Bone (PTB) and any of the following: radiographic (X-ray, Magnetic Resonance Imaging (MRI), or bone scan) or evidence of bone necrosis
* The subject has an Ankle-Brachial Index ≥ 0.7 to ≤ 1.3 or TcPO2 ≥ 40 mmHg on the dorsum of the affected foot, or Great Toe Pressure ≥ 50 mmHg
* The subject is under the care of a physician for the management of Diabetes Mellitus
* The subject is willing to return for all mandatory visits as defined in the protocol
* The subject is willing to follow the instructions of the trial Investigator

Exclusion Criteria:

* The subject's index ulcer is primarily located on the dorsal surface of the foot
* The subject's index ulcer can be addressed by primary closure through the completion of the initial or staged surgical procedure
* The subject has a contralateral major amputation of the lower extremity
* The subject has a glycated hemoglobin A1c (HbA1c) level of > 12% †
* The subject has been on oral steroid use of > 7.5 mg daily for greater than seven (7) consecutive days in 30 days before Screening
* The subject has been on parenteral corticosteroids, or any cytotoxic agents for seven consecutive days in the period of 30 days before Screening
* The subject is currently taking the type 2 diabetes medicine canagliflozin (Invokana™, Invokamet™, Invokamet XR™)
* The subject has malignancy or a history of cancer, other than non-melanoma skin cancer, in five years before Screening
* The subject is pregnant
* The subject is a nursing mother
* The subject is a woman of child-bearing potential who is unwilling to avoid pregnancy or use an appropriate form of birth control (adequate birth control methods are defined as: topical, oral, implantable, or injectable contraceptives; spermicide in conjunction with a barrier such as a condom or diaphragm; intrauterine contraceptive device; or surgical sterilization of partner).
* The subject is unable to sustain off-loading as defined by the protocol
* The subject has an allergy to primary or secondary dressing materials used in this trial
* The subject has an allergy to glycerol
* The subject's index ulcer is over an acute Charcot deformity
* The subject has had previous use of NEOX®, CLARIX®, or TTAX01 applied to the index ulcer
* Per Investigator's discretion the subject is not appropriate for inclusion in the trial, e.g., undergoing surgical treatments listed in the protocol or the subject currently has sepsis, i.e., life-threatening organ dysfunction caused by a dysregulated host response to infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Complete wound healing | over 25 weeks
  Time from baseline to initial observation of healing, where healing has been confirmed at two consecutive visits each two weeks apart.

SECONDARY OUTCOMES:
Wound durability | by Week 26
  Proportion of wounds that re-ulcerate
Limb preservation | by Week 26
  proportion of minor and major amputations following the initial procedure
Patient-reported mobility | Baseline to End of Study (approximately 26 weeks)
  compare total score on PROMIS Health Organization Neuro-QoL 'lower extremity function'; scale from 1-5; higher scores indicate better self-reported health

CONTACTS AND LOCATIONS:
Overall Officials: Seema Kumbhat, MD, Study Chair — Chief Medical Officer
Locations (16):
- United States (16):
  - LakeView Clinical Research, Guntersville, Alabama
  - Banner University Medical Center Tucson, Tucson, Arizona
  - Clemente Clinical Research, Los Angeles, California
  - VA Northern California Health Care System, Mather, California
  - CureCentric, Palmdale, California
  - PIH Health, Whittier, California
  - Midland Florida Clinical Research Center, DeLand, Florida
  - Delray Physician Care Center, Delray Beach, Florida
  - Gateway Clinical Trials, LLC, O'Fallon, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Reno Orthopedic Clinic, Reno, Nevada
  - Curalta Foot and Ankle, Westwood, New Jersey
  - Cutting Edge Research, LLC, Circleville, Ohio
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Advantage Foot Care of Houston, Houston, Texas
  - Biolife Genetics Research, Houston, Texas

IPD SHARING:
Plan to Share IPD: No